CLINICAL TRIAL: NCT06939907
Title: Clinical Trial to Evaluate the Efficacy and Safety of Nexpowder™ for Diverticular Bleeding in the Lower Gastrointestinal Tract: A Prospective, Multi-Center, Single-Arm, Open-Label, Pilot Clinical Trial
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Nexpowder™ for Diverticular Bleeding in the Lower Gastrointestinal Tract
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nexpowder_008
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Lower Gastrointestinal Bleeding; Diverticular Bleeding
MeSH Terms: conditions — Diverticular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nexpowder Treatment Arm (Experimental)
  Interventions: Device: Nexpowder™

INTERVENTIONS:
Device: Nexpowder™ — Nexpowder™ hemostatic powder

SUMMARY:
Clinical Trial to Evaluate the Efficacy and Safety of Nexpowder™ for Diverticular Bleeding in the Lower Gastrointestinal Tract

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older at the time of screening
* Patients diagnosed with diverticular bleeding

Exclusion Criteria:

* Patients diagnosed with upper gastrointestinal bleeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate | 30 days post treatment
  30 days after successful endoscopic hemostasis

SECONDARY OUTCOMES:
Hemostasis rate | Immediately after the procedure
  Hemostasis rate
Rebleeding rate | 7 days post treatment
  Rebleeding rate

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - Chosun University Hospital, Gwangju
  - Sejong Chungnam National University Hospital, Sejong
  - Kangdong Kyunghee University Hospital, Seoul
  - Yangsan Busan National University Hospital, Yangsan